CLINICAL TRIAL: NCT05814237
Title: Perpetual Observational Study of Acute Respiratory Infections Presenting Via Emergency Rooms and Other Acute Hospital Care Settings
Brief Title: POS-ARI-ER Observational Study of Acute Respiratory Infections
Acronym: POS-ARI-ER
Status: Recruiting | Type: Observational
Sponsor: European Clinical Research Alliance for Infectious Diseases (ECRAID) (Other)
Collaborators: UMC Utrecht (Other); University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: ECRAID-Base POS-ARI-ER
Record Dates: First submitted 2023-02-27; First posted 2023-04-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Respiratory Infection; Acute Respiratory Tract Infection
Keywords: Infections; Communicable Diseases
MeSH Terms: conditions — Infections; Communicable Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasal and throat swab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — Data collection from study participants to characterise diagnostic and therapeutic practices.

SUMMARY:
Acute respiratory infections (ARI) are one of the most frequent reasons for hospital admission and antibiotic use, and can be caused by a broad range of pathogens, including respiratory viruses with proven epidemic potential, e.g. influenza and coronaviruses. The POS-ARI-ER study will focus on describing the different routine diagnostic and therapeutic practices in the work-up and treatment of ARI, as well as clinical outcomes across the patient population. In addition, POS-ARI-ER aims to characterise both the adult patient population with ARI presenting to acute hospital settings in Europe, and the aetiology of ARI in these patients.

DETAILED DESCRIPTION:
The POS-ARI-ER study is a perpetual, observational study (POS), designed to provide data for clinical characterisation of acute respiratory infections (ARIs) in adults presenting to hospital settings across Europe.

Establishing the etiological cause of ARI at the time of presentation is difficult with currently available diagnostic approaches. Improvements in diagnosis and strategies for use of targeted antibiotic and antiviral treatment strategies are needed to improve patient outcomes, and to reduce selection of antimicrobial resistance (AMR) and antiviral resistance. Recent advances in routine diagnostics in secondary care settings include molecular tests that can detect multiple pathogens simultaneously, and highly sensitive and specific point of care tests that can provide attending clinicians with rapid results. However, the implementation of these technologies into routine clinical practice within hospitals, and any impact on treatment decisions or patient outcomes, has not been widely evaluated.

The aim is to accurately characterise cases of ARIs presenting to acute hospital services, such as emergency departments and acute medical assessment units, in Europe.

Characterisation will focus on identifying the routine diagnostic methods (laboratory and point of care testing) and pharmacological interventions employed by different centres in patients presenting with ARI. Data will be collected using standardised report forms that capture clinical, laboratory and prescribing information. Participants will include those who require admission to hospital, as well as patients who are discharged the same day from the emergency department or acute medical assessment unit. In addition, a subset of participants will have single upper respiratory tract research sample (e.g. nose/throat swab) obtained at enrolment (within 24 hours), for pathogen detection by molecular methods.

Describing the variations in routine practice provides a foundation both to improve patient care through currently available approaches, as well as to inform areas of focus for development of new strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical suspicion of a new episode of acute respiratory tract infection, with onset in the last 10 days
* Patient presents to an emergency room or secondary care setting
* Informed consent is provided by patient or their legal representative

Exclusion Criteria:

* Patient has been transferred from another hospital
* Patient admitted to hospital for >2 days at the time of enrolment
* Patient has been previously enrolled in the POS-ARI-ER study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with community acquired acute respiratory infections presenting to acute hospital settings in Europe.
Sampling Method: Non-Probability Sample
Enrollment: 11750 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of adult patients undergoing ARI-relevant microbiology and virology investigations. | Four years
  Calculate the proportion of types of ARI-relevant microbiology and virology investigations performed.
Proportion of adult patients receiving antibiotics, antivirals, antifungals and/or immunomodulators. | Four years
  Calculate the proportion of cases receiving antibiotics, antivirals, antifungals and/or immunomodulators.
Clinical outcome of adults with community acquired ARI in acute hospital settings in Europe. | Last day in hospital, at death or 28 days after admission, whichever comes first.
  Maximal score using the ordinal scale assessed at discharge, death or at 28 days after hospital admission: 6= death, 5= hospitalisation requiring extracorporeal membrane oxygenation (ECMO) and/or invasive mechanical ventilation, 4= hospitalisation requiring non invasive ventilation (NIV) and/or high flow nasal cannula (HFNC) oxygen therapy, 3= requiring supplemental oxygen (but not NIV/HFNC), 2= hospitalisation not requiring supplemental oxygen, 1= not hospitalised.
Length of hospital and/or ICU stay in adults with community acquired ARI in acute hospital settings in Europe. | Last day in hospital, at death or 28 days after admission, whichever comes first.
  Number of days patient admitted to hospital or ICU.
Duration of NIV and IMV/ECMO in adults with community acquired ARI in acute hospital settings in Europe. | Last day in hospital, at death or 28 days after admission, whichever comes first.
  Number of days patients receiving NIV and IMV/ECMO.
All cause mortality in adults with community acquired ARI in acute hospital settings in Europe. | Last day in hospital, at death or 28 days after admission, whichever comes first.
  Total number of deaths for each ARI-related pathogen.

SECONDARY OUTCOMES:
Patient demographics of the adult patient population with ARI presenting to acute hospital settings in Europe. | Four years
  Evaluate demographics of patient population with ARI.
Comorbidities in the adult patient population with ARI presenting to acute hospital settings in Europe. | Four years
  Evaluation of comorbidities in patient population with ARI.
Presenting symptoms in the adult patient population with ARI presenting to acute hospital settings in Europe. | Four years
  Evaluation of presenting symptoms in the adult patient population with ARI.
Physiological measurements in the adult patient population with ARI presenting to acute hospital settings in Europe. | Four years
  Evaluation of the physiological measurements in the adult patient population with ARI.
Aetiology of ARI in adults presenting to acute hospital settings in Europe. | Four years
  Detection of putative pathogens in respiratory tract samples (research upper respiratory tract sample at presentation and ARI-relevant microbiology/virology results obtained through routine clinical care).

OTHER OUTCOMES:
Association between clinical outcomes and diagnostic or treatment related variables, for different aetiologies of community acquired ARI in adults presenting to hospital across Europe. | Last day in hospital, at death or 28 days after admission, whichever comes first.
  Maximal score on ordinal scale assessed at discharge, death or at 28 days after hospital admission: 6= death, 5= hospitalisation requiring extracorporeal membrane oxygenation (ECMO) and/or invasive mechanical ventilation, 4= hospitalisation requiring non invasive ventilation (NIV) and/or high flow nasal cannula (HFNC) oxygen therapy, 3= requiring supplemental oxygen (but not NIV/HFNC), 2= hospitalisation not requiring supplemental oxygen, 1= not hospitalised, stratified by pathogen.

CONTACTS AND LOCATIONS:
Locations (23):
- Erasme Hospital, Brussels, Belgium
- University Hospital for Infectious Diseases, Zagreb, Zagreb, Croatia
- France (4):
  - CHU Grenoble, Grenoble
  - CHU Limoges, Limoges
  - CHU Lyon, Lyon
  - CHU de Tours, Tours
- General University Hospital of Patras, Pátrai, Greece
- Azienda Ospedaliera Policlinico di Bari, Bari, Italy
- Netherlands (2):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Radboud University Medical Center, Nijmegen
- Romania (3):
  - Agrippa Ionescu Hospital, Carol Davila University of Medicine and Pharmacy Bucharest, Bucharest
  - Infectious and Tropical Diseases Hospital "Dr. Victor Babes", Bucharest
  - Cluj Napoca Infectious Disease Clinical Hospital, Cluj-Napoca
- General Hospital, Kragujevac, Kragujevac, Serbia
- Spain (2):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Virgen Macarena, Seville
- United Kingdom (7):
  - Craigavon Area Hospital, Craigavon
  - NHS Lothian- Royal Infirmary of Edinburgh and St Johns Hospital, Edinburgh
  - Gateshead Health NHS Foundation Trust, Gateshead
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Royal Free London NHS Foundation Trust - Royal Free Hospital, London
  - Sheffield Teaching Hospitals NSH Foundation Trust, Sheffield
  - South Tyneside and Sunderland NHS Foundation, Sunderland

IPD SHARING:
Plan to Share IPD: No